CLINICAL TRIAL: NCT04969744
Title: Impact of Cold Exposure on Metabolic Regulation in Children With Non Alcoholic Fatty Liver Disease (NAFLD)
Acronym: ICE BAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); Guts UK (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 278804
Record Dates: First submitted 2021-06-23; First posted 2021-07-21 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: ICE BAT study will be performed in two stages. In stage 1, we will recruit 12 to 24 healthy volunteers aged between 16-26 years.
  In stage 2, we will recruit 12 children aged between 8-16 years with NAFLD and 12 age- and sex-matched controls (healthy volunteers).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intermittent Cold Exposure (ICE) (Experimental): Stage 1- healthy volunteers aged 16-26 years will receive ICE for one day. stage 2a - controls aged 8-16 will receive ICE for one day. Stage 2b- NAFLD patients aged 8-16 years will receive ICE for one day or choose to continue for 5 days.
  Interventions: Device: ICE

INTERVENTIONS:
Device: ICE — Intermittent Cooling Exposure using cooling garment for 1-2 hours

SUMMARY:
The aim of this project is to generate pilot data for a grant proposal to evaluate the impact of intermittent cold exposure (ICE) on brown and white adipose tissue (BAT/WAT) function in children with non-alcoholic fatty liver disease (NAFLD). The condition NAFLD is the most common liver disease in both adults and children. There are many emerging drug therapies for NAFLD but at considerable cost in terms of potential side effects. In a mouse model of diet-induced obesity, ICE was shown to help activate BAT, which may help NAFLD and other obesity associated health risks. Given that children have more BAT than adults, we hypothesise that intermittent cold exposure via a cooling vest in children with NAFLD will increase BAT stores or function. We will investigate whether intermittent cold exposure via a cooling vest device will stimulate BAT and also establish whether the cooling vest is acceptable to children and young people. If it is acceptable and has an impact on BAT function this could be a new treatment to reduce the severity of metabolic disorders associated with obesity, particularly fatty liver, e.g. hepatic steatosis. In stage 1, we will investigate the impact of intermittent cold exposure (ICE) on brown and white adipose tissue (BAT/WAT) function in young people aged 16 to 26 years old, as a feasibility study to optimise the cooling process. In stage 2, we will investigate the impact of ICE on BAT and WAT function in 8-16 year olds with non-alcoholic fatty liver disease (NAFLD) and matched controls. Participants will have thermal imaging, MRI scans and provide samples before and after wearing the cooling vest.

DETAILED DESCRIPTION:
ICE BAT is a single centre pilot study.

In stage 1, 12 to 24 young people aged 16-26 will be recruited into the study. Participants will use a cooling garment (for 1-2 hours). MRI scans and thermal imaging will be performed before and after ICE to evaluate BAT size and activation. Liver steatosis will be evaluated using MRI Proton Dense Fat Fraction (PDFF). Serum markers of BAT activation and glucose/lipid metabolism will be measured before and after ICE.

In stage 2,12 children with NAFLD and 12 age- and sex-matched controls will be enrolled in the study. In stage 2a, healthy controls will use a cooling garment (for 1-2 hours) and undergo MRI scan and thermal imaging before and after ICE to evaluate BAT size and activation. Liver steatosis will be evaluated using MRI PDFF. In stage 2b the NAFLD patients will be asked to attend for one day and if they are happy to continue, will use a cooling garment (for 1-2 hours/day for a further 4 days). MRI scans and thermal imaging will be performed before and after ICE on day 1 and day 5 to evaluate BAT size and activation. Liver steatosis will be evaluated using MRI PDFF. Serum markers of BAT activation and glucose/lipid metabolism will be measured on day 1 and day 5. Participants with NAFLD, will be asked to give a faecal sample for analysis of their gut microbiome before the study and after day 5 of ICE treatment.

ELIGIBILITY:
Inclusion Criteria:

Stage 1: Young Adult 16-26 year olds

* Individual must be aged 16-26 years
* Individual who has voluntarily signed informed consent

Stage 2: Children 8-16 year olds

* Child aged 8-16 years old with NAFLD attending the paediatric clinic at Kings College Hospital
* A control group of children with a BMI z score <1.5 and no diagnosis of liver disease
* Individual willing to participate in the study with informed consent. If the participant is under 16, the parent should provide informed consent.

Exclusion Criteria:

Stage 1: Young Adult 16-26 year olds

* Individual who is thought to be too unwell to participate by the study team, e.g. if participant has a fever or infection requiring treatment with antibiotics.
* Individual who has a medical condition that requires treatment with a drug that could alter BAT function, e.g. thyroid disease (thyroxine, carbimazole, propylthiouracil, beta- blockers), liver disease (ursodeoxycholic acid), any condition requiring treatment with peroxisome proliferator-activated receptor gamma (PPAR-γ) agonists or 4 beta 3 adrenoceptor (β3-AR) agonists.
* Individual has smoked/vaped 5 days before participating in the study.

Stage 2: Children 8-16 year olds

* Participant who is thought to be too unwell to participate by the study team, e.g. if participant has a fever or infection requiring treatment with antibiotics.
* Individual who has a medical condition that requires treatment with a drug that could alter BAT function, e.g. thyroid disease (thyroxine, carbimazole, propylthiouracil, beta- blockers), liver disease (ursodeoxycholic acid), any condition requiring treatment with peroxisome proliferator-activated receptor gamma (PPAR-γ) agonists or 4 beta 3 adrenoceptor (β3-AR) agonists
* Individual has smoked/vaped 5 days before participating in the study

Ages: 8 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-10-23 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Effectiveness in participants aged 16-26 | One day
  Assess the ability to deliver ICE via a cooling garment using a probe to measure skin temperature at regular intervals during ICE treatment.
Stage 1: Acceptability in participants aged 16-26 | One day
  Acceptability will be measured by the sum of participants' responses to questions 1-5 of the questionnaire. Responses to individual items will also be presented.
Stage 2: Effectiveness for 8-16 year old participants. | One to Five days
  Assess the ability of ICE to deliver cooling, using a probe to measure skin temperature at regular intervals during ICE treatment.
Stage 2: Acceptability for 8-16 year old participants. | One to Five days
  Acceptability of the cooling jacket will be measured by the sum of participants' responses to questions 1-5 of the questionnaire. Responses to individual items will also be presented. Patients will be given the choice as to whether they are willing to attend for 5 days and undergo a further MRI, thermal imaging and blood sampling on day 5.

SECONDARY OUTCOMES:
Stage 1: BAT dimensions: Measured using MRI before and after ICE. | One Day
  Measurement of brown adipose tissue depots will be recorded using MRI scans before and after ICE.
Stage 1: BAT and WAT function: Assessed using MRI measurements before and after ICE. | One Day
  Using measures of blood flow, fat fraction and water fraction taken during MRI, analysis analysis algorithms are used to distinguish between BAT and WAT, with blood flow measurements used as a surrogate marker of BAT function.
Stage1 : BAT activity: Measured using thermal imaging before and after ICE. | One Day
  Thermal imaging will be analysed for average temperature of the BAT region of interest and the upper chest area before and after ICE treatment.
Stage 1: Acceptability of study protocol and cooling garment: Measured using an acceptability questionnaire at the end of the study. | One Day
  As above
Stage 1: Autonomic function measured by the Empatica E4 device for the duration of the study. | One Day
  As above
Stage 1: Dietary information: Assessed using a 24 hour dietary recall at the beginning of the study day 1. | One Day
  As above
Stage1: Lipid profile: Measured through analysis of blood spot (collected before and after ICE, mandatory) by a secondary laboratory. | One Day
  As above
Stage1: Glucose measured before and after ICE (mandatory). | One Day
  Glucose measured (in mmol/l) before and after ICE.
Stage1: Metabolic hormone profile: Measured before and after ICE (optional). | One Day
  Metabolic hormones measured before and after ICE, on serum samples by research laboratory.
Stage1: Serum lipids measured before and after ICE (optional). | One Day
  Serum lipids measured before and after ICE (optional) through Viapath Laboratory, King's College Hospital.
Stage 2: BAT dimensions measured using MRI before and after ICE. | One to Five days
  Measurement of brown adipose tissue depots will be recorded using MRI scans before and after ICE, on day 1 for stage 2a and day 1 and day 5 for stage 2b participants.
Stage 2: BAT and WAT function assessed using MRI measurements before and after ICE. | One to Five days
  Using measures of blood flow, fat fraction and water fraction taken during MRI, analysis analysis algorithms are used to distinguish between BAT and WAT, with blood flow measurements used as a surrogate marker of BAT function.
Stage 2: Liver fat fraction(proton dense fat fraction (PDFF)): Measured in percentage using MRI before ICE on day 1 for stage 2a and before ICE on day 1 and after ICE on day 5 for stage 2b (PDFF measured using MRI). | One to Five days
  As above
Stage 2: BAT activity: Measured using thermal imaging before and after ICE on day 1 for stage 2a and day 1 and day 5 for stage 2b participants. | One to Five days
  As above
Stage 2: Acceptability of study protocol and cooling garment. | One to Five days
  Measure using an acceptability questionnaire at the end of the study. The willingness of the participants to attend for 5 days is also a reflection on the acceptability of the study.
Stage 2: Autonomic function measured by the Empatica E4 device. | One to Five days
  As above
Stage 2: Activity measured using the Fitbit for NAFLD patients completing 5 days of ICE. | One to Five days
  As above
Stage 2: Dietary information: Assessed using a 24 hour dietary recall, completed at the beginning of study day 1 (and on Day 5 for NAFLD patients who continue to five days). | One to Five days
  As above
Stage 2: Lipid profile: Measured through analysis of blood spot (collected before and after ICE on day 1 for stage 2a and day 1 and day 5 for stage 2b, mandatory) by an external laboratory. | One to Five days
  As above.
Stage 2: Serum lipid measurements before and after ICE (optional) | One to Five days
  Serum lipids measured before and after ICE (optional) through Viapath Laboratory, King's College Hospital.
Stage 2: Metabolic hormone profile before and after ICE (optional). | One to Five days
  Metabolic hormones measured before and after ICE, on serum samples by research laboratory.
Stage 2: Glucose measurements before and after ICE in stage 2 participants | One to Five days
  Glucose measurements before and after ICE in mmol/l.
Stage 2: Gut microbiome evaluation in NAFLD participants (optional). | One to Five days
  Bacterial DNA will be isolated from faecal samples to study 16S RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Ovadia, Doctor, Principal Investigator — King's College London
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
N/A - no plan to share identifiable patient data with other researchers.